CLINICAL TRIAL: NCT04151784
Title: Factors That Impact the Relationship Between Pulmonary Status and Susceptibility to Electronic Cigarette Use
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohammed Alqahtani, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300003376
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Electronic Cigarette Use; Pulmonary Disease
Keywords: Susceptibility to Electronic Cigarette Use
MeSH Terms: conditions — Vaping; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Group: Pulmonary Group who have evidence of pulmonary diseases
  Interventions: Other: Pulmonary Group
- Healthy Control: Health Group who have no evidence of pulmonary diseases
  Interventions: Other: Healthy Control

INTERVENTIONS:
Other: Pulmonary Group — Data collection will be obtained on the day an individual has an appointment at the pulmonary clinic. After patients meet with their pulmonary physicians, the physicians will inform them about the study and explain that participation is voluntary. If a patient agrees, the researcher will provide copies of the questionnaires and again clarify that participation is voluntary. The workflow of the clinic will not be interrupted while the researcher conducts the study, and he will only ask participants to fill out the questionnaires if they have enough time to participate.
  Groups: Pulmonary Group
Other: Healthy Control — The second group will be recruited as a control group consisting of healthy adult participants through purposive convenience sampling at other collaborating UAB sites. The principal investigator will collect self-report responses through a questionnaire packet given to anyone willing to participate in the study
  Groups: Healthy Control

SUMMARY:
The purpose of the study is to explores various psycho-social, physiological, cognitive, behavioral, and environmental factors that may affect the association between pulmonary status and Susceptibility to Electronic Cigarette Use

DETAILED DESCRIPTION:
In this study self-report questionnaires will be distributed and it should take between 20-25 minutes. Participants will be be asked questions related to smoking history, e-cigarette use, psychosocial factors, behavioral factors, environmental factors, and cognitive factors.

There is also an option of taking a web-based survey, Qualtrics® (Qualtrics, Provo, UT), if they do not have enough time to complete the surveys at this time. The online version of the questionnaires will be sent to the one week from now.

There is also a follow-up 5 minutes call with 6 months after today to follow-up with any change regarding to e-cigarette use.

ELIGIBILITY:
Inclusion Criteria:

Pulmonary Are 18 years of age or older. Attend outpatient Pulmonary clinic at UAB Diagnosed with a pulmonary disease Speak English as primary language Are medically stable and without psychiatric disorders. Signed Informed consent Healthy Are 18 years of age or older. Free from any pulmonary disease Report good to excellent general health Speak English as primary language Signed Informed consent

Exclusion Criteria:

Pulmonary Are younger than 18 years of age Do not attend the outpatient pulmonary clinic at UAB (pulmonary group) Report current e-cigarette use Are non-English speakers Have unstable medical or psychiatric disorders as determined by the assigned medical doctor (pulmonary group) Refuse to sign the informed consent

Healthy Are younger than 18 years of age Report any pulmonary diseases (control group) Report fair to poor general health (control group) Report current e-cigarette use Are non-English speakers Refuse to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort will be divided into two groups according to their pulmonary status: subjects who are diagnosed with any pulmonary disease (pulmonary group) and those without any pulmonary disease (control group).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
To examine psychosocial (stress, depression, anxiety) as mediators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  The DASS-21 is a clinical assessment that measures the state of depression, It has 21 questions. The internal consistency of the DASS-21 scales was acceptable (depression: alpha = .829). The scale range is from 0 to 28 + with 0 being closest to normal and 28+ being extremely severe. The DASS-21 is a clinical assessment that measures the state of anxiety, It has 21 questions. The internal consistency of the DASS-21 scales was acceptable (anxiety : alpha = .778). The scale range is from 0 to 20 + with 0 being closest to normal and 20+ being extremely severe. The DASS-21 is a clinical assessment that measures the state of stress, It has 21 questions. The internal consistency of the DASS-21 scales was acceptable (stress : alpha = .871). The scale range is from 0 to 37 + with 0 being closest to normal and 37+ being extremely severe
To examine physiological variables (quality of life) as mediators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  The Health Survey SF-12 questionnaire will be used to assess the quality of life (Ware, Kosinski, & Keller, 1996). The SF-12 is a reliable and valid instrument. Internal consistency, test-retest reliability, construct (convergent and discriminant) validity, and criterion (concurrent and predictive) validity have been shown to be adequate (continuous variable). The minimum score is 0 and maximum score is 100, and higher scores mean a better quality of life and lower score mean worse outcome.
To examine physiological variables (Respiratory Symptoms) as mediators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  Questions that was developed by (Leidy, 2003) will be used to assess Breathlessness, Cough, Sputum, and chest tightness. Each symptom will be tested individually for its mediating effect, and they will be combined as one composite score to test the total mediating effect. The minimum score is 0 and maximum score is 25, and higher scores mean a worse respiratory symptoms and lower score mean better respiratory symptoms.
To examine physiological variables (Eating Disorder Questionnaire) as mediators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  12 questions adopted from Gideon et al. (2016) will be used to discover which participants believe that they suffer from eating disorders. This measure showed high internal consistency (Cronbach's α = .913) and temporal stability (ICC = .93; p < .001) (continuous variable). These range from a score of zero ("no symptoms") to three ("extreme symptoms").
To examine cognitive variables (Belief) as mediators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  A short form of the e-cigarette consequence questionnaire will be used to assess the e-cigarette expectancy questionnaire. This questionnaire was developed and validated by Peter S. Hendricks et al. (2014). Cronbach's alpha reliabilities of the e-cigarette-specific range from .67 to .88 (ordinal variable). This questionnaire has 25 statements. Each statement contains a possible consequence of smoking an e-cigarette. For each of the statements, participants should rate how LIKELY or UNLIKELY that they believe each consequence is for them when they use an e-cigarette. If the consequence seems LIKELY to them, they should circle a number from 5-9. That is, if they believe that a consequence would never happen, circle 0; if they believe a consequence would happen every time they smoke, circle 9. If it seems a little unlikely to them, they would circle 4
To examine cognitive variables (Risk Perception) as mediators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  Questions that have been successfully used in previous studies (Adkison et al., 2013; Choi & Forster, 2013; Nicksic et al., 2017; Stein et al., 2015) will be used to assess the participants' risk perception of e-cigarettes (ordinal variable). There are six statements that assess the participants' perception toward e-cigarette, and the participants should choose between 1 to 5 where 1 means "strongly disagree" and 5 means "strongly agree".
To examine cognitive variables (attitudes toward e-cigarettes) as mediators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  The Comparing E-cigarettes and Cigarettes Questionnaire (CEAC) will be used to assess attitudes towards e-cigarettes compared to cigarettes. The CEAC is a 17-item self-report measure with three factors: (1) General Benefits (seven items; α = 0.85), (2) Addiction/Cessation Benefits (five items; α = 0.89), and (3) Improve Health (five items; α = 0.92) (Hershberger, Karyadi, VanderVeen, & Cyders, 2017). The CEAC has been shown to be positively related to e-cig use (b 0.41-1.24, p < .01) and has demonstrated good psychometric properties (α 0.83-0.93) (ordinal variable). There are ten statements that assess the participants' perception toward e-cigarette, and the participants should choose between 1 to 5 where 1 means "strongly disagree" and 5 means "strongly agree".
To examine cognitive variables (intention to quit) as mediators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  A scale of 1 to 10 has been used before by Peter S. Hendricks et al. (2014) will be used to assess the desire to quit smoking and the success of quitting among smokers (continuous variable). (Scale of 1 to 10 with 1 = No desire to quit and 10 = full desire to quit).
To examine behavioral variables (Alcohol And Drug Use) as moderators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  They will be assessed using a previously used questionnaire (P. S. Hendricks, Delucchi, Humfleet, & Hall, 2012) (categorical variable). Participants should choose "Yes" or "No" based to see if they drink alcohol or use any of the addictive substance.
To examine environmental variables (Advertisement) as moderators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  To assess different areas related to some environmental factors, the following questions will be asked: "When you are using the Internet, how often do you see ads or promotions for e-cigarettes," "When you read newspapers or magazines, how often do you see ads or promotions for e-cigarettes," "When you go to a convenience store, supermarket, or gas station, how often do you see ads or promotions for e-cigarettes," and "When you watch TV, how often do you see ads or promotions for e-cigarettes." Participants can choose from a Likert scale with responses range from 1 to 6 where 1 means ("No use/watch/see/go") and 6 means "always". This question has been successfully used in previous Centers for Disease Control and Prevention (CDC) studies (ordinal variable).
To examine environmental variables (Warning Labels) as moderators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  To assess awareness of warning labels on e-cigarettes and associated paraphernalia, we will use the following question: "During the past 30 days, how often did you see a warning label on an e-cigarette package?" Participants can choose from 6 Likert scale categories in order for them to answer the preceding questions. 1 indicates "I did not see an e-cigarette package during the past 30 days" and 6 indicates always. This question has been successfully used in previous Centers for Disease Control and Prevention (CDC) studies (ordinal variable).
To examine environmental variables (Exposure to Special Prices ) as moderators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  Exposure to special price offers for e-cigarettes will be assessed by asking: "In the last 30 days, have you noticed any special price offers, such as discounts or coupons, for e-cigarettes/vaping devices or e-liquid?" Response options include "Yes" and "No". This question has been successfully used in previous Centers for Disease Control and Prevention (CDC) studies (categorical variable).
To examine environmental variables (Exposure to E-cigarette Vapors from Some in An indoor or Outdoor Public Place ) as moderators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  A question will be asked regarding number of days that someone breathes vapor from someone who was using an e-cigarette in an indoor or outdoor public place. This question has been successfully used in previous Centers for Disease Control and Prevention (CDC) studies (continuous variable).
To examine environmental variables (Using E-cigarettes in Home) as moderators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  The following question will be asked regarding using e-cigarettes in home "Does anyone who lives with you use e-cigarette?" (yes/no). This question has been successfully used in previous Centers for Disease Control and Prevention (CDC) studies (categorical variable).
To examine environmental variables (suggestion to Use E-cigarettes by Healthcare Provider) as moderators of the relationship between pulmonary disease status and susceptibility to using e-cigarettes. | Through study completion, an average of 1 year
  A question will be asked to see if e-cigarette use was suggested by a healthcare provider. This question has been successfully used by Harrington et al. (2014) in previous studies (yes/no) (categorical variable).
Susceptibility to e-cigarette use | Through study completion, an average of 1 year
  The questionnaire that will be used in our study was adopted from a study performed by Nicksic, Snell, Rudy, Cobb and Barnes (44). Nicksic, Snell, Rudy, Cobb and Barnes (44) adapted a validated measure on susceptibility to smoking. The adapted survey scale for measuring susceptibility to using e-cigarette showed a high degree of internal consistency (Cronbach's alpha = 0.97). The susceptibility to e-cigarette use score is constructed based on participants' responses to the following questions: (1) Do you think that you will use an e- cigarette soon? (2) Do you think that in the future you might experiment with e-cigarettes? (3) Do you think you will use an e-cigarette in the next year? and (4) If one of your best friends were to offer you an e-cigarette, would you smoke it? After each question, participants could endorse "Definitely not," "Probably not," "Probably yes," and "Definitely yes." (Continuous variables).
Nicotine addiction as a moderating variable between pulmonary status and the e-cigarette use. | Through study completion, an average of 1 year
  The Penn State Cigarette Dependence Index (PS-CDI) to assess cigarette dependence. The PS-CDI (α = .72) both have fair to good internal consistency (Foulds et al., 2015). The PS-CDI also appears to be a valid measure of the dependence construct, capturing self-perceived addiction, heavy use, early use after overnight deprivation, and continued use over time (continuous variable). The Penn State Cigarette Dependence Index (PS-CDI) to assess cigarette dependence. The PS-CDI (α = .72) both have fair to good internal consistency (Foulds et al., 2015). The PS-CDI also appears to be a valid measure of the dependence construct, capturing self-perceived addiction, heavy use, early use after overnight deprivation, and continued use over time (continuous variable). Scoring: 0-3= not dependent, 4-8 low dependence, 9-12 medium dependence, 13+ = high dependence

SECONDARY OUTCOMES:
Demographic variables | Through study completion, an average of 1 year
  Demographic information will be collected from participants by using questions adopted from the National Adult Tobacco Survey Questionnaire. Different question will be used about gender, age, income, and education.
Health information | Through study completion, an average of 1 year
  The following question will be used to assess participants' health status: "In general, how is your health?" (Excellent, very good, good, fair, poor). This question has been successfully used in previous studies
Pulmonary Status | Through study completion, an average of 1 year
  ICD-10-CM (International Classification of pulmonary diseases) will be used to determine if the healthy adults have a history of pulmonary disease.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined

REFERENCES:
- [Derived] Alqahtani MM Jr, Alanazi AMM, Aljohani H, Ismaeil TT, Algarni SS, Alotaibi TF, Alotaibi MM, Kalan ME, Lein DH, Alqahtani MK, Alwadeai KS, Almutairi AB, Hendricks PS. The relationship between chronic lung disease diagnosis and the susceptibility to e-cigarette use in adults: The mediation effects of psychosocial, cognitive influences, and the moderation effect of physiological factors. Tob Induc Dis. 2023 Sep 22;21:116. doi: 10.18332/tid/169741. eCollection 2023. PMID 37745030